CLINICAL TRIAL: NCT01612104
Title: Psychological First Aid With Children in a High Risk Group - a Repeated Single Case Design
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NORCE Norwegian Research Centre AS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RKBU62
Record Dates: First submitted 2012-05-31; First posted 2012-06-05 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Post Traumatic Stress Disorder; Adjustment Disorder
Keywords: Post Traumatic Stress Disorder; Anxiety symptoms; Depressive symptoms; Externalizing behavior; Reduced quality of life
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Adjustment Disorders; Anxiety Disorders; Depression | interventions — Psychological First Aid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Psychological First Aid (Experimental): Psychological material developed for children and adolescents, based on cognitive behavioral theory, used to structure therapeutic conversations and/or for self-help.
  Interventions: Behavioral: Psychological First Aid

INTERVENTIONS:
Behavioral: Psychological First Aid — A cognitive behavioral (CBT) method structuring and focusing psychological therapy sessions with children and adolescents having been exposed to potential trauma

SUMMARY:
The purpose of this pilot-study is to evaluate a cognitive behavioral method "Psychological First Aid" used with a group of children (11-16 years) in high risk of developing psychological problems. Participants are recruited from a low-threshold program ("The Children's House in Oslo") where counseling is given to children suspected of being physically or sexually abused, or having witnessed domestic violence. The study includes twelve children and teenagers that receive 2 to 6 sessions of counseling. Psychological problems (e.g. anxiety, depression, reactions to trauma) and quality of life will be assessed at pre- post and follow-up (after 3, 6 and 12 months). In addition, some symptoms of will be assessed daily.

ELIGIBILITY:
Inclusion Criteria:

* Children/adolescents that:

  * contact "The Children's House in Oslo" after having experienced potential traumatic event(s).
  * are assessed as having psychological symptoms related to potential trauma
  * are between 11 and 16 years old
  * agree to participate in the study (both the youth and his/her parents(s)
* understand and speak Norwegian

Exclusion Criteria:

- Children/adolescents with:

* mental retardation
* reading skills below 8 year
* psychosis
* high risk of suicidal behavior is assumed

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2012-03; Primary Completion 2013-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Children's Revised Impact of Event Scale (CRIES) | One year

SECONDARY OUTCOMES:
Child Post-Traumatic Cognition Inventory (CPTCI) | One year

CONTACTS AND LOCATIONS:
Overall Officials: Bente SM Haugland, PhD, Principal Investigator — Centre for Child and Adolescent Mental Health, Western Norway
Locations (1):
- The Children's House in Oslo, Oslo, Norway